CLINICAL TRIAL: NCT06827093
Title: Augmented Dyadic Interventions to Boost Quality of Life Among Stroke Survivors and Care Partners in Pakistan.
Brief Title: Dyadic Interventions to Boost Quality of Life Among Stroke Survivors and Care Partners in Pakistan.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Nazia Shuaib, Principal Investigator, Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-135; NBC-R NO,4-87/NBC-839/23/762 (Other: National bioethical committee for research(NBC-R))
Record Dates: First submitted 2024-08-12; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Stroke
Keywords: Stroke survivor; Dyadic intervention

STUDY DESIGN:
Intervention Model Description: single-blind, randomized controlled trials with repeated measures
Who Masked: Participant
Masking Description: single-blind, randomized controlled trials with repeated measures, The primary investigator trained two qualified nurses in each province continuously for 2 weeks to deliver interventions to promote fairness. Permission was obtained from the tertiary care hospital to check the medical records of the study population and to contact them based on their medical records after 2 weeks of discharge. First, the patients were contacted by telephone for inclusion criteria based on their records and being voluntary participants in the study, and then pretest data was collected. The experimental group were received five sessions, while the control group ere received only routine care. The first post-test was conducted three months after the intervention, the second post-test was conducted six months later, and the third post-test was conducted 12 months later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This program's protocol will consist of Part I (three structured in-person education sessions) and Part II (two telephone follow-up sessions). The session and content of the intervention will be:
  Session 1 (Two weeks after discharge) Introduction to stroke and different aspects of management: Session 2 (three weeks after discharge)
  Promotion of care and demonstration of self-care activities:
  Demonstration and skill development Session 3 (Four weeks after discharge) Psychological adjustment and management: Session 4 (2 weeks later from 3rd session) Telephonic session: The aim of communicating with the dyad through the telephone is to provide the information required for psychological support, behavioural regulation and emotional support.
  Session 5 (2 weeks later from 3rd session) Followup telephonic session: Promoting activities and assistance
  Interventions: Other: Skill Building Dyadic Intervention
- Controlled group (Other): While the control group will receive their routine care. The first post-test will be conducted three months after the intervention, the second post-test will be conducted six months later, and the third post-test will be conducted 12 months later. The inclusion and exclusion criteria for the patient and caregiver will be the same.
  Interventions: Other: Skill Building Dyadic Intervention

INTERVENTIONS:
Other: Skill Building Dyadic Intervention — The focal point of skill-building interventions contains some strategies that facilitate problem-solving, goal setting, communicating with care experts, stress management, hands-on training in such skills (lifting and mobility techniques and assistance with activities of daily living), and modification of communication according to the needs of stroke survivors.

SUMMARY:
This study (RCTs) will be conducted on stroke survivors and their care partners after discharge from the hospital. The study will aim to evaluate the impact of augmented dyadic intervention on the quality of life of stroke survivors and caregiver burden. A randomized control trial with a parallel group design will be used for the study. The design used for the current study will be single-blind, randomized controlled trials with repeated measures. Each group will include 196 subjects (98 stroke survivors and 98 care partners). The total number of individuals will be 392, including 196 stroke survivors and 196 care partners. Stroke survivors will have an age range of 18-75 years and both genders with a confirmed diagnosis of stroke. The goal of this study will be to rehabilitate patients with disability, there is a dire need for dyad interventions to support and train stroke care partners by providing education, counselling, emotional support and access to health services. The hypothesis of this (RCTs )is that there is no relationship between stress and quality of life for improvement in quality of life through dyadic intervention.

DETAILED DESCRIPTION:
Stroke is a leading cause of mortality and disability around the world, leaving survivors with significant physical deficits and resulting in a variety of psychological problems as well as social constraints and retreats for both the survivors and their families. The study population will be stroke survivors and their care partners after discharge from the hospital. The design will be single-blind, randomized controlled trials with repeated measures. A total of 392 participants will be recruited voluntarily, of which 196 will be randomly assigned to the control group and 196 to the intervention group. A five-session intervention containing three face-to-face and two telephonic sessions will be delivered. A valid and reliable stroke-specific quality of life questionnaire for stroke survivors and Zarit Burden and an interview for caregiver burden will be used. The primary investigator will train two qualified nurses in each province for 2 weeks to deliver interventions to promote fairness. Permission will be obtained from the tertiary care hospital to check the medical records for the study population and to contact them based on their medical records after 2 weeks of discharge. First, the patients will be contacted by telephone for inclusion criteria based on their records and being voluntary participants in the study, and then pretest data will be collected. The experimental group will receive five sessions, while the control group will receive routine care. The first post-test will be conducted three months after the intervention, the second post-test will be conducted six months later, and the third post-test will be conducted 12 months later Data analysis will be performed through SPSS 22 as descriptive (frequency and percentages for categorical variables, while the mean and standard deviation for continuous variables) and inferential statistics (independent t-test for differences between the groups and Pearson correlation for association with demographic variables).

ELIGIBILITY:
Inclusion Criteria:

* The study includes stroke survivors:

  * Having an age range of 18-75 years with a confirmed diagnosis of stroke (confirmed by a neurologist with radiological evidence by either CT scan and/or MRI) and meeting the following eligibility criteria was required. 26
  * Having a diagnosis of stroke More than 15 days
  * Stable, non-fluctuating stroke with no acute, ongoing neurological
  * No preexisting disability before stroke (defined by mRS =0).
  * Independent in daily living activities before the stroke
  * Expected to return home with residual disability

While the inclusion criteria for care partners was an identified primary care partner greater than 18 years of age,

1. Able to speak
2. Urdu speaker
3. Care partners include aphasic patients and demented patients.
4. No significant physical or psychological disability
5. Be willing and able to provide support to patients after discharge

Exclusion Criteria: Exclusion criteria for stroke survivors

1. Acute illness (i.e., dementia, advanced cancer, hepatic or renal failure or fractured lower extremity)
2. Preexisting diseases before stroke
3. Life expectancy of 6 months or less.
4. Post-invasive procedural strokes like CABG, angiography and post-operative stroke
5. Global aphasia and/or being unable to communicate. Dementia on the Mini-Mental State Examination (of <22) (due to inability to directly communicate) 26,27
6. History of ongoing psychoactive substance abuse, terminal illnesses like renal failure or end-stage cancer
7. The presence of psychiatric morbidity before and after stroke, which specifically includes manic disorders, schizophrenia

Exclusion criteria for family caregivers

1. having an age greater than 80 years 2. Acute illness

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
promoting the quality of life and care of stroke patients | 12 months of intervention
  This study will evaluate the effects of a skill-building dyadic intervention on improving the quality of life (QOL) for 392 individuals, consisting of 196 stroke survivors and their 196 care partners. The study will utilize a 49-item stroke-specific questionnaire to assess the quality of life of stroke survivors across 12 domains. This comprehensive tool will provide valuable insights into the various aspects of stroke survivors' lives. The study's outcome is expected to reveal significant improvements in the quality of life of stroke survivors. After receiving the intervention, participants will report enhanced knowledge, satisfaction, and self-efficacy. Specifically, the study will find positive impacts on energy, mobility, mood, and treatment efficacy, ultimately leading to an improved quality of life for stroke survivors.

SECONDARY OUTCOMES:
Reduces the burden of dyad members | 12 months
  The Zarit Burden Interview (ZBI) will assess caregiver burden using a modified 22-item scale. This scale will feature a 5-point Likert scale (0-4) across four domains: confidence, competence, quality of care, and self-efficacy. Data analysis will utilize Pearson correlation through SPSS 26.0 to explore the relationship between stroke survivors and caregiver burden with demographic variables. This study aims to reduce stroke survivors' and caregivers' psychological, social, and financial burdens. A single-blind, randomized controlled trial with 392 participants (196 stroke survivors, 196 care partners) will test a 5-session intervention, with data collection at pre-intervention, and post-intervention (3, 6, 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Nazia Shuaib, PhD, Principal Investigator — Zhengzhou University Henan China
Locations (1):
- Dr.Nazia, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data (IPD) from this clinical trial to facilitate further research and transparency."Individual participant data (IPD) will be shared upon request, following publication of primary results, through a secure online platform, with terms outlined in a data use agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within 6 to 12 months after completion of my study
Access Criteria: IPD will be shared upon request, within 6 to 12 months of publication

REFERENCES:
- [Background] Arntzen C, Borg T, Hamran T. Long-term recovery trajectory after stroke: an ongoing negotiation between body, participation and self. Disabil Rehabil. 2015;37(18):1626-34. doi: 10.3109/09638288.2014.972590. Epub 2014 Oct 16. PMID 25318537
- [Background] Pucciarelli G, Ausili D, Rebora P, Arisido MW, Simeone S, Alvaro R, Vellone E. Formal and informal care after stroke: A longitudinal analysis of survivors' post rehabilitation hospital discharge. J Adv Nurs. 2019 Nov;75(11):2495-2505. doi: 10.1111/jan.13998. Epub 2019 Apr 22. PMID 30883880
- [Background] Dharma KK, Damhudi D, Yardes N, Haeriyanto S. Increase in the functional capacity and quality of life among stroke patients by family caregiver empowerment program based on adaptation model. Int J Nurs Sci. 2018 Sep 7;5(4):357-364. doi: 10.1016/j.ijnss.2018.09.002. eCollection 2018 Oct 10. PMID 31406848
- [Background] McCurley JL, Funes CJ, Zale EL, Lin A, Jacobo M, Jacobs JM, Salgueiro D, Tehan T, Rosand J, Vranceanu AM. Preventing Chronic Emotional Distress in Stroke Survivors and Their Informal Caregivers. Neurocrit Care. 2019 Jun;30(3):581-589. doi: 10.1007/s12028-018-0641-6. PMID 30421266
- [Background] Shaffer KM, Riklin E, Jacobs JM, Rosand J, Vranceanu AM. Mindfulness and Coping Are Inversely Related to Psychiatric Symptoms in Patients and Informal Caregivers in the Neuroscience ICU: Implications for Clinical Care. Crit Care Med. 2016 Nov;44(11):2028-2036. doi: 10.1097/CCM.0000000000001855. PMID 27513536
- [Background] Pucciarelli G, Ausili D, Galbussera AA, Rebora P, Savini S, Simeone S, Alvaro R, Vellone E. Quality of life, anxiety, depression and burden among stroke caregivers: A longitudinal, observational multicentre study. J Adv Nurs. 2018 Apr 27. doi: 10.1111/jan.13695. Online ahead of print. PMID 29700840
- [Background] Shyu YI, Maa SH, Chen ST, Chen MC. Quality of life among older stroke patients in Taiwan during the first year after discharge. J Clin Nurs. 2009 Aug;18(16):2320-8. doi: 10.1111/j.1365-2702.2008.02458.x. Epub 2008 Sep 17. PMID 18800991
- [Background] Catangui EJ, Slark J. Nurse-led ward rounds: a valuable contribution to acute stroke care. Br J Nurs. 2012 Jul 12-25;21(13):801-5. doi: 10.12968/bjon.2012.21.13.801. PMID 22874780
- [Background] Javier Catangui E, John Roberts C. The lived experiences of nurses in one hyper-acute stroke unit. Br J Nurs. 2014 Feb 13-26;23(3):143-8. doi: 10.12968/bjon.2014.23.3.143. PMID 24526021
- [Background] Mou H, Lam SKK, Chien WT. Effects of a family-focused dyadic psychoeducational intervention for stroke survivors and their family caregivers: a pilot study. BMC Nurs. 2022 Dec 21;21(1):364. doi: 10.1186/s12912-022-01145-0. PMID 36544154
- [Background] Ostwald SK, Godwin KM, Cron SG, Kelley CP, Hersch G, Davis S. Home-based psychoeducational and mailed information programs for stroke-caregiving dyads post-discharge: a randomized trial. Disabil Rehabil. 2014;36(1):55-62. doi: 10.3109/09638288.2013.777806. Epub 2013 Apr 17. PMID 23594060
- [Background] Krishnan S, Pappadis MR, Weller SC, Fisher SR, Hay CC, Reistetter TA. Patient-centered mobility outcome preferences according to individuals with stroke and caregivers: a qualitative analysis. Disabil Rehabil. 2018 Jun;40(12):1401-1409. doi: 10.1080/09638288.2017.1297855. Epub 2017 Mar 21. PMID 28320217
- [Background] Deyhoul N, Vasli P, Rohani C, Shakeri N, Hosseini M. The effect of family-centered empowerment program on the family caregiver burden and the activities of daily living of Iranian patients with stroke: a randomized controlled trial study. Aging Clin Exp Res. 2020 Jul;32(7):1343-1352. doi: 10.1007/s40520-019-01321-4. Epub 2019 Aug 31. PMID 31473982
- [Background] Cheng HY, Chair SY, Chau JPC. Effectiveness of a strength-oriented psychoeducation on caregiving competence, problem-solving abilities, psychosocial outcomes and physical health among family caregiver of stroke survivors: A randomised controlled trial. Int J Nurs Stud. 2018 Nov;87:84-93. doi: 10.1016/j.ijnurstu.2018.07.005. Epub 2018 Jul 28. PMID 30059815
- [Background] Tang SH, Chio OI, Chang LH, Mao HF, Chen LH, Yip PK, Hwang JP. Caregiver active participation in psychoeducational intervention improved caregiving skills and competency. Geriatr Gerontol Int. 2018 May;18(5):750-757. doi: 10.1111/ggi.13246. Epub 2018 Jan 22. PMID 29356339

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT06827093/Prot_SAP_ICF_000.pdf